CLINICAL TRIAL: NCT01374256
Title: Effectiveness of Imipenem and Sulbactam in the Treatment of Bacteremic Patients Contracted With Imipenem-resistant Acinetobacter Baumannii
Brief Title: Imipenem and Sulbactam in the Treatment of Imipenem-resistant Acinetobacter Baumannii Bacteremia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Te-li Chen, MD, PhD, Associate Professor, Division of Infectious Diseases, Department of Medicine, Taipei Veterans General Hospital
Other Study IDs: ISP 38889; 201012032ID (Other: IRB of Taipei Veterans General Hospital)
Record Dates: First submitted 2011-06-14; First posted 2011-06-15 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: Acinetobacter Bacteraemia
Keywords: carbapenem; sulbactam; Acinetobacter baumannii

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Acinetobacter baumannii isolates from the blood samples of patients
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Combination therapy: Patients with Acinetobacter baumannii bacteremia treated with combination therapy of imipenem and sulbactam
- Not combination therapy: Patients with Acinetobacter baumannii bacteremia not treated with combination therapy of imipenem and sulbactam

SUMMARY:
Infections caused by imipenem-resistant Acinetobacter baumannii are associated with high mortality and morbidity. The treatment choices for this resistant pathogen are limited.

The objective of the present proposal is to evaluate the effectiveness of combination therapy of imipenem and sulbactam in patients contracted with A. baumannii, and to correlate the clinical effect with the in vitro synergistic results.

DETAILED DESCRIPTION:
Acinetobacter baumannii has been increasingly reported in the outbreak of nosocomial infections in the intensive care units, which not only prolong the length of hospital stay but result in high attributable mortality. With its intrinsic resistance to many antimicrobial agents and rapid acquirement of resistance mechanism, resistance to carbapenems, which is often accompanied with resistance to multiple drugs, has emerged worldwide. The limited treatment choice included tigecycline, colistin, and sulbactam. However, the low serum level and bacteriostatic nature of tigecycline hamper its application in blood stream infection, one of the most common presentations of A. baumannii infections. The nephrotoxicity and neurotoxicity of intravenous colistin have caused great concerns in critically ill patients whereas immediate bronchospasm after inhalation and significant clinical consequences have been reported. Sulbactam has been used for decades in combination of ampicillin and well tolerated. However, the emergence of resistance strains and discourage of monotherapy in severely ill patients make combination an attractive choice. Combination of sulbactam and carbapenems has good synergism against A. baumannii with elevated minimal inhibitory concentration (MIC) of sulbactam and/or carbapenems while in an animal model using A. baumannii with higher MIC of both sulbactam and meropenem, survival rate was higher in combination group than sulbactam or meropenem-treated alone group. The similar in vivo bactericidal effect was also observed in combination of imipenem and sulbactam. Despite plenty of in vivo and in vitro studies mentioned above, the clinical studies were limited. Besides, the information regarding the correlation of in vitro synergistic effect of carbapenem and sulbactam with the clinical effect is rarely mentioned. Therefore, our study is aimed to evaluate the effectiveness of combination therapy of imipenem and sulbactam in patients contracted with A. baumannii, and to correlate the clinical effect with the in vitro synergistic results

ELIGIBILITY:
Inclusion Criteria:

* elder than 18 years old are included if they have bloodstream infections due to A. baumannii regardless of primary infection sites

Exclusion Criteria:

* pregnancy or lactation in women
* history of serious allergy or intolerance to study drug therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study will be conducted at Taipei Veterans General Hospital, a 2900-bed tertiary care medical center in Taiwan. Patients elder than 18 years old are included if they have bloodstream infections due to A. baumannii regardless of primary infection sites.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
survival rate | 14 days

SECONDARY OUTCOMES:
survival rate | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Te-Li Chen, PhD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taiwan, Taipei, Taiwan, Taiwan